CLINICAL TRIAL: NCT06712914
Title: Rapid Non-Invasive Brain Stimulation for Hoarding Disorder
Acronym: TMS-HOLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77098
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hoarding Disorder; Hoarding; Clutter
Keywords: TMS; hoarding disorder; hoarding; clutter; iTBS
MeSH Terms: conditions — Hoarding Disorder; Hoarding; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Theta-burst stimulation (TBS) (Experimental): Theta-burst stimulation (a form of transcranial magnetic stimulation) targeting the right frontal pole.
  Interventions: Device: MagPro X100 by MagVenture

INTERVENTIONS:
Device: MagPro X100 by MagVenture — Participants will receive 5 session per day of TBS for 6 days (30 sessions total). Six treatment days have to occur within a 2 week period. Each session will be comprised of 1800 pulses, using a MagVenture MagPro X100.

SUMMARY:
This study explores whether rapid non-invasive brain stimulation can help reduce hoarding disorder symptoms.

DETAILED DESCRIPTION:
Hoarding disorder (HD) is characterized by difficulty letting go of possessions, leading to clutter that congests living spaces and impairs daily functioning. The majority of HD patients treated with cognitive behavioral therapy for HD usually experience considerable residual symptoms. New treatments are greatly needed. This study explores whether rapid non-invasive brain stimulation can help reduce hoarding disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Primary diagnosis of hoarding disorder
3. Sufficient severity of hoarding symptoms
4. Willing and able to understand and complete consent and study procedures

Exclusion Criteria:

1. Psychiatric or medical conditions or medications that make participation unsafe
2. Pregnant or nursing females
3. Previous exposure to TMS or ECT
4. History of any implanted device or psychosurgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Compulsive Acquisition Scale (CAS) | Change from baseline to 3 weeks after treatment starts
  The Compulsive Acquisition Scale (CAS) is an 18-item questionnaire that measures the extent to which individuals acquire and feel compelled to acquire possessions.
  The total score (sum of 18 items) ranges from 0 to 126. Total score higher than 48 shows significant difficulty with acquiring.

OTHER OUTCOMES:
Change in Hoarding Symptom Severity as Measured by Saving Inventory-Revised (SI-R) | Change from baseline to 3 weeks after treatment starts
  The Saving Inventory-Revised scale (SI-R) is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.
  The total score (sum of 23 items) ranges from 0 to 92. Total score higher than 41 shows significant difficulty with clutter.
  For the acquisition subscale, items 2 (reverse score), 9, 11, 14, 16, 18 and 21 are summed together. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with excessive acquisition.
  For the difficulty discarding subscale, items 4(reverse score), 6, 7, 13, 17, 19, 23 are summed together. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with discarding.
  For the clutter subscale, items 1, 3, 5, 8, 10, 12, 15, 20, 22 are summed together. The subscale ranges from 0 to 36 and score greater than 15 indicates difficulty with accumulated clutter.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rodriguez Lab Website — https://med.stanford.edu/rodriguezlab/home.html
- See also: Dr. Carolyn Rodriguez (PI) Stanford Faculty Profile — https://med.stanford.edu/profiles/carolyn-rodriguez?tab=bio